CLINICAL TRIAL: NCT07366710
Title: Quantification of Amino Acid and Glucose Metabolism in Healthy Controls and Patients With Non-alcoholic Fatty Liver Disease Using Total- Body PET
Brief Title: Measuring Amino Acid and Glucose Metabolism in Healthy Volunteers and NAFLD Patients Using Total-body PET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Per Cramon, Physician, Rigshospitalet, Denmark
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 565_23
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Glucose Metabolism; NAFLD (Nonalcoholic Fatty Liver Disease)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Fluorodeoxyglucose F18; (18F)fluoroethyltyrosine; Glucagon; Somatostatin; Sodium Chloride; Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy Controls: FDG (oral & IV) (Experimental): Healthy volunteers receive 18F-FDG by oral administration and intravenous administration on separate study days, including an oral glucose tolerance test visit. Total-body PET/CT imaging is performed after each tracer administration.
  Interventions: Drug: 18F-FDG (oral); Drug: 18F-FDG (intravenous); Other: Oral Glucose Tolerance Test
- Healthy Controls: FET (oral & IV) (Experimental): Healthy volunteers receive 18F-FET by oral administration and intravenous administration on separate study days. Dynamic and static total-body PET/CT imaging is performed.
  Interventions: Drug: 18F-FET (oral); Drug: 18F-FET (intravenous)
- Healthy Controls: Oral FET + Glucagon/Somatostatin Clamp (Crossover) (Experimental): Healthy participants undergo two study days with oral ^18F-FET administration combined with either glucagon infusion during a pancreatic clamp (somatostatin infusion) or placebo. Total-body PET/CT imaging is performed using a crossover design.
  Interventions: Drug: 18F-FET (oral); Drug: Glucagon; Drug: Somatostatin; Drug: Sodium chloride (placebo)
- NAFLD Patients: Oral FET + Glucagon/Somatostatin Clamp (Crossover) (Experimental): Participants with NAFLD undergo two study days with oral ^18F-FET administration combined with either glucagon infusion during a pancreatic clamp (somatostatin infusion) or placebo. Total-body PET/CT imaging is performed using a crossover design.
  Interventions: Drug: 18F-FET (oral); Drug: Glucagon; Drug: Somatostatin; Drug: Sodium chloride (placebo)

INTERVENTIONS:
Drug: 18F-FDG (oral) — Oral administration of 18F-fluorodeoxyglucose (^18F-FDG) for total-body PET/CT to assess gastrointestinal absorption, systemic biodistribution, and whole-body glucose metabolism.
  Arms: Healthy Controls: FDG (oral & IV)
Drug: 18F-FDG (intravenous) — Intravenous bolus administration of 18F-fluorodeoxyglucose (18F-FDG) for total-body PET/CT to measure systemic biodistribution and whole-body glucose metabolism.
  Arms: Healthy Controls: FDG (oral & IV)
Drug: 18F-FET (oral) — Oral administration of O-(2-[18F]fluoroethyl)-L-tyrosine (18F-FET) for total-body PET/CT to assess gastrointestinal amino acid absorption and whole-body amino acid metabolism.
  Arms: Healthy Controls: FET (oral & IV); Healthy Controls: Oral FET + Glucagon/Somatostatin Clamp (Crossover); NAFLD Patients: Oral FET + Glucagon/Somatostatin Clamp (Crossover)
Drug: 18F-FET (intravenous) — Intravenous bolus administration of O-(2-[18F]fluoroethyl)-L-tyrosine (18F-FET) for total-body PET/CT to measure systemic amino acid biodistribution and dynamic metabolic kinetics.
  Arms: Healthy Controls: FET (oral & IV)
Drug: Glucagon — Continuous intravenous glucagon infusion to stimulate hepatic amino acid metabolism during a pancreatic clamp.
  Arms: Healthy Controls: Oral FET + Glucagon/Somatostatin Clamp (Crossover); NAFLD Patients: Oral FET + Glucagon/Somatostatin Clamp (Crossover)
Drug: Somatostatin — Continuous intravenous somatostatin infusion to suppress endogenous pancreatic hormone secretion during the pancreatic clamp.
  Arms: Healthy Controls: Oral FET + Glucagon/Somatostatin Clamp (Crossover); NAFLD Patients: Oral FET + Glucagon/Somatostatin Clamp (Crossover)
Drug: Sodium chloride (placebo) — Intravenous infusion of isotonic sodium chloride solution used as placebo during crossover comparison with glucagon infusion.
  Arms: Healthy Controls: Oral FET + Glucagon/Somatostatin Clamp (Crossover); NAFLD Patients: Oral FET + Glucagon/Somatostatin Clamp (Crossover)
Other: Oral Glucose Tolerance Test — Standard oral glucose load (75 g in 250 mL water) to assess glucose-stimulated metabolic responses during PET/CT.
  Arms: Healthy Controls: FDG (oral & IV)

SUMMARY:
This observational study aims to quantify whole-body amino acid and glucose metabolism in healthy adults and in patients with non-alcoholic fatty liver disease (NAFLD) using total-body PET/CT. The study investigates how orally and intravenously administered PET tracers (18F-FDG and 18F-FET) are absorbed in the gastrointestinal tract, distributed across major organs, and metabolized in different physiological and pathological states. A further objective is to examine how glucagon, during a pancreatic clamp using somatostatin, influences amino acid metabolism in healthy individuals and whether this response is altered in patients with NAFLD.

Participants will be healthy volunteers or patients with NAFLD, aged 18-70 years. Depending on study group, participants will undergo one or more total-body PET/CT scans following oral or intravenous tracer administration, and in some cases receive glucagon or placebo infusion. Blood samples will be collected during scanning to assess hormone levels and metabolic responses. Data from these imaging sessions will be used to characterize nutrient metabolism, compare oral and intravenous tracer kinetics, and explore glucagon-induced metabolic changes across study groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Body mass index (BMI) 20-27 kg/m2

Exclusion Criteria:

* Pregnancy
* Claustrophobia
* Inability to give consent due to psychological or other causes
* Inability to speak/read Danish
* Diabetes, cancer (active or treated within the last five years) or inflammatory diseases.
* Low albumin
* Chronic disorders that require medical treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Whole-body tracer uptake (SUVmean) assessed using total-body PET/CT | 0-180 minutes after tracer administration

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen University Hospital - Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No